CLINICAL TRIAL: NCT01843920
Title: A Prospective, Randomized Study Comparing the Effects of Topical Aqueous Suppressants on Intraocular Gas Duration Following Scleral Buckling and Pneumatic Retinopexy.
Brief Title: The Effect of Glaucoma Drops on of the Duration of a Pure Intraocular Gas Bubble
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Hsu, MD (Other)
Responsible Party: Sponsor-Investigator, Jason Hsu, MD, Investigator, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11095 Gas Duration; 11-095 (Other: Wills Eye IRB)
Record Dates: First submitted 2013-04-18; First posted 2013-05-01 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Scleral Buckling
Keywords: eye; pneumatic retinopexy; topical
MeSH Terms: interventions — dorzolamide-timolol combination; dorzolamide; Standard of Care; Adrenal Cortex Hormones; Prednisolone; Polymyxin B; Trimethoprim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post surgery without glaucoma drops (Active Comparator): This will be for the group that had gas duration surgery using SF6 (Sulfur Hexafluoride) or C3F8 (perfluoropropane gas tamponade) and only uses the standard post-operative topical drops.
  Interventions: Drug: standard post-operative topical drops
- Post surgery with glaucoma drops (Experimental): This will be for the group that had gas duration surgery (using SF6 or C3F8). In addition to the standard post-operative topical drops, glaucoma drops, Timolol-dorzolamide (timolol 0.5%-dorzolamide 2%) will be given.
  Interventions: Drug: Timolol-dorzolamide (Glaucoma drops); Drug: standard post-operative topical drops

INTERVENTIONS:
Drug: Timolol-dorzolamide (Glaucoma drops) — Patients will receive the standard post-operative drops regardless of what group you are in. The glaucoma drops will only be given to the experimental group.
  Other Names: timol; glaucoma drops; dorzolamide; timol-dorzolamide
  Arms: Post surgery with glaucoma drops
Drug: standard post-operative topical drops — Patients will receive the standard post-operative drops regardless of what group ther are in. The standard post-operative drops are Prednisolone acetate,Polymyxin B and Trimethoprim
  Other Names: glaucoma; drops; standard of care; oral; corticosteroid; prednisolone; Polymyxin B; trimethoprim

SUMMARY:
A controlled clinical study comparing the effect of topical aqueous suppressants on intraocular gas duration.

DETAILED DESCRIPTION:
A Prospective, Randomized Study Comparing the Effects of Topical Aqueous Suppressants on Intraocular Gas Duration following Scleral Buckling and Pneumatic Retinopexy

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Have undergone eye surgery including scleral buckling or pneumatic retinopexy for treatment of retinal detachment other condition at the discretion of the investigator.

Exclusion Criteria:

* Prior surgery to treat glaucoma.
* Current use of glaucoma eye drops.
* Absence of a lens in the eye or presence of a lens implant in front of the iris (colored part of your eye).
* Allergy or contraindication to any of the glaucoma drops being used in this study (e.g., sulfa allergy, asthma, chronic obstructive pulmonary disease (bronchitis or emphysema), slow heart rate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post Surgery Without Glaucoma Drops | Post Surgery With Glaucoma Drops
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post Surgery Without Glaucoma Drops | Post Surgery With Glaucoma Drops | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Resolution of Intraocular Gas Bubble
Description: This will be reported by the patient when they see/feel the gas bubble disappear.
Time Frame: Following surgery, until gas bubble is gone. Up to 2 months.
Measure: Mean (Full Range); unit: Duration in days, gas bubble
Arm/Group | Post Surgery Without Glaucoma Drops | Post Surgery With Glaucoma Drops
Number analyzed (Participants) | 12 | 9
Duration in days, gas bubble | 40.4 [27 to 51] | 37.8 [29 to 50]

2. Secondary Outcome: Number of Participants With Return of Intraocular Pressure to Normal Levels
Description: Number of participants with a normal intraocular pressure of 10-21 mm Hg at the Month 2 visit
Time Frame: Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | Post Surgery Without Glaucoma Drops | Post Surgery With Glaucoma Drops
Number analyzed (Participants) | 12 | 9
Participants
  High IOP at Month 2 | 1 | 0
  Normal IOP at Month 2 | 7 | 7
  Low IOP at Month 2 | 1 | 0
  Data Not Available | 3 | 2

ADVERSE EVENTS:
Arm/Group | Post Surgery Without Glaucoma Drops | Post Surgery With Glaucoma Drops
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes